CLINICAL TRIAL: NCT07381907
Title: Effects of Transcranial Direct Current Stimulation Over the Supplementary Motor Area Combined With Nordic Walking on Gait and Balance in Parkinson's Disease
Brief Title: Effects of Transcranial Direct Current Stimulation Combined With Nordic Walking on Gait and Balance in Parkinson's Disease
Acronym: tDCS+NW-PD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Luciane Lobato Sobral, Principal Investigator, Universidade Metodista de Piracicaba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UEPA-PD-SMA-001; CAAE: 86894625.0.0000.8767 (Other: CONEP/Plataforma Brasil (CEP))
Record Dates: First submitted 2026-01-19; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Parkinson Disease (PD); Gait Disorders; Postural Balance
Keywords: transcranial direct current stimulation; nordic walking; parkinson disease; gait; postural balance; motor cortex; rehabilitation
MeSH Terms: conditions — Parkinson Disease; Mobility Limitation | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Parallel assignment with two arms (1:1): (i) active anodal tDCS over the supplementary motor area delivered concurrently with standardized Nordic Walking, and (ii) sham tDCS with the same Nordic Walking protocol. Randomization uses computer-generated permuted blocks; allocation is concealed with sequentially numbered, opaque, sealed envelopes prepared by an independent researcher. Participants receive 12 sessions over 4 weeks (3×/week).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, treating therapists and outcome assesors are blinded. The stimulator is pre-programmed under coded modes so that active and sham display identical indicators; sham includes brief ramp-in/out to mimic sensations then no sustained current. Session procedures and Nordic Walking are identical across arms to preserve blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS over SMA + standardized Nordic Walking (Experimental): Participants receive anodal tDCS over the supplementary motor area (SMA) delivered concurrently with a standardized 30-minute Nordic Walking (NW) session, 3×/week for 4 weeks (12 sessions). tDCS: 2.0 mA, 20 min, saline-soaked sponge electrodes (5×7 cm), anode over midline SMA (FCz), cathode supraorbital contralateral; 30-s ramp-in/out. NW protocol identical across both arms (warm-up, technique practice with poles, continuous walking at moderate effort, cool-down).
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS), active; Behavioral: Standardized Nordic Walking program
- Sham tDCS + standardized Nordic Walking (Sham Comparator): Participants undergo the same NW protocol (30 min) on the same schedule (3×/week for 4 weeks; 12 sessions) while receiving sham tDCS with brief ramp-in/out to mimic sensations and no sustained current; electrodes and device indicators match the active condition.
  Interventions: Device: Sham transcranial Direct Current Stimulation; Behavioral: Standardized Nordic Walking program

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS), active — Anodal tDCS over SMA (FCz) with saline-soaked sponge electrodes (5×7 cm); cathode supraorbital contralateral; 2.0 mA for 20 minutes, 30-s ramp-in/out; delivered during NW; 12 sessions over 4 weeks (3×/week).
  Arms: Active tDCS over SMA + standardized Nordic Walking
Device: Sham transcranial Direct Current Stimulation — Same montage and timing as active; brief ramp-in/out then 0 mA for the remainder; delivered during NW; 12 sessions over 4 weeks.
  Arms: Sham tDCS + standardized Nordic Walking
Behavioral: Standardized Nordic Walking program — 30-minute supervised session (5-min warm-up; 20-min continuous walking with poles at moderate perceived exertion; 5-min cool-down); technique cues for pole use and cadence; performed each visit in both arms; 12 sessions over 4 weeks.

SUMMARY:
Parkinson's disease can cause slow or unsteady walking and balance problems that raise the risk of falls. This study will test whether adding a gentle, non-invasive brain stimulation called transcranial direct current stimulation (tDCS) during a supervised Nordic Walking program improves mobility in people with Parkinson's disease. Participants will be randomly assigned to receive either active tDCS or an inactive (sham) procedure that feels the same but does not deliver current, while both groups complete the same supervised walking program. Sessions occur three times per week for four weeks. We will measure walking speed with a 10-Meter Walk Test as the main outcome, and also evaluate balance, motor symptoms, quality of life, and any side effects. We expect that tDCS given during the walking sessions will help people walk faster and feel steadier compared with the walking program alone.

DETAILED DESCRIPTION:
Parkinson's disease (PD) commonly presents with gait slowing, reduced step length, balance impairment and freezing of gait, leading to falls and loss of independence. The supplementary motor area (SMA) is a key hub for internally generated movement, sequencing, and gait initiation. Anodal transcranial direct current stimulation (tDCS) over SMA can increase cortical excitability and modulate cortico-basal ganglia networks. Nordic Walking (NW) is a task-specific, cue-rich gait training method that promotes rhythmic arm-leg coupling, stride elongation, and postural control. Delivering SMA-targeted tDCS concurrently with NW is expected to leverage state-dependent plasticity, priming motor networks while patients practice the target skill, thereby enhancing the functional yield of training.

Objectives and hypotheses: The primary objective is to determine whether anodal SMA tDCS given during NW improves walking speed more than sham tDCS during the same NW program. We hypothesize superiority of the active condition on gait speed (10-Meter Walk Test) at post-intervention, with maintenance at 1-month follow-up. Secondary objectives include effects on balance, motor signs, and disease-specific quality of life, and documentation of safety/tolerability.

Design and setting: Single-center, parallel-group, randomized, double-blind, sham-controlled clinical trial conducted at a university outpatient neurorehabilitation facility in Brazil. Participants are randomized 1:1 using a computer-generated sequence (permuted blocks) by an investigator not involved in enrollment or assessments. Allocation is concealed using sequentially numbered, opaque, sealed envelopes stored in a secure location accessible only to the randomization custodian. Masking and fidelity: Participants, treating therapists, and outcome assessors remain blinded. The stimulator is pre-programmed under coded modes; device indicators and procedures are identical across groups. The sham program includes brief current ramp-in/out to mimic sensations, then no sustained current. Intervention fidelity is supported by standardized checklists, session logs, and periodic supervision of therapists not involved in outcome assessment. Participants: Adults with idiopathic PD on stable antiparkinsonian medication who can follow simple commands. The sample targets a slow-gait phenotype to maximize clinical relevance. Exclusion criteria address contraindications to tDCS (e.g., implanted cranial/brain devices, non-intact scalp at electrode sites), unsafe exercise participation, cognitive impairment incompatible with consent/testing, and concurrent neuromodulation trials. Assessments are scheduled in a standardized medication state (e.g., "on" medication) to reduce variability. Interventions: Active tDCS + NW - Anodal tDCS over SMA (midline, approximately FCz) using saline-soaked sponge electrodes (5×7 cm); cathode supraorbital contralateral. Intensity 2.0 mA for 20 minutes with 30-s ramp-in/out, three sessions/week for 4 weeks (12 sessions). Stimulation is delivered concurrently with NW. The NW session lasts 30 minutes (5-min warm-up; 20-min continuous walking with poles at moderate effort monitored by perceived exertion; 5-min cool-down), supervised by trained staff with standardized instruction on pole technique and cadence. Sham tDCS + NW - Identical setup, timing, and NW protocol; sham involves brief ramping then zero current for the remainder of the stimulation window. Other therapies and exercises are not allowed during the trial. Outcomes and assessment schedule: The primary outcome is gait speed (m/s) on the 10-Meter Walk Test at post-intervention and 1-month follow-up, referenced to baseline. Secondary outcomes include Timed Up and Go, Berg Balance Scale, Freezing of Gait Questionnaire, MDS-UPDRS Part III, and PDQ-39; adverse events are recorded each session using a structured checklist. Assessments occur at baseline, post-intervention, and 1-month follow-up under standardized conditions and assessor training. Sample size and statistical analysis: The trial is powered to detect a between-group difference in gait speed consistent with a minimally important change in PD, allowing for attrition. The primary analysis uses ANCOVA with post-intervention gait speed as the dependent variable, group as fixed effect, and baseline gait speed as covariate; corresponding estimates with 95% confidence intervals and effect sizes are reported. Sensitivity analyses include linear mixed-effects models across baseline, post, and follow-up time points. Analyses follow the intention-to-treat principle with appropriate handling of missing data (e.g., maximum likelihood/multiple imputation); a per-protocol analysis is planned as supportive. Responder analyses (e.g., proportion achieving ≥0.10 m/s improvement) and exploratory subgroup analyses (e.g., disease severity, baseline freezing status) are prespecified. Safety and monitoring: Vital signs (heart rate, blood pressure, SpO₂) are checked pre/post sessions; skin under electrodes is inspected before/after stimulation. Common tDCS sensations (tingling, itching, mild erythema) and exercise-related symptoms are systematically queried. Predefined criteria permit pausing or discontinuation (e.g., severe headache, dizziness, hypertensive response, arrhythmia, significant skin irritation). Serious adverse events are reported promptly to the ethics board per institutional policy. Data management and dissemination: De-identified data are stored on secure, access-controlled servers with audit trails; only authorized study personnel can access the linkage file. Results will be disseminated through peer-reviewed publications and scientific meetings. Individual-participant data sharing will adhere to the plan stated in the IPD section of this record.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease (e.g., UK Brain Bank criteria)
* Hoehn & Yahr stage II-IV (on medication)
* Stable antiparkinsonian medication for ≥4 weeks before enrollment
* Slowed gait phenotype (e.g., ≥6 seconds on 10-Meter Walk at preferred speed)
* Able to ambulate at least 10 meters with or without a cane/poles (no hands-on assistance from a therapist)
* Able to follow simple commands; provides written informed consent (MMSE ≥24 or equivalent cognitive screening)
* Willing to maintain stable PD medication and usual care during the 4-week intervention, unless medically required

Exclusion Criteria:

* Contraindications to tDCS: implanted cranial/brain devices (e.g., DBS), metal in the skull (excluding dental), active skin disease/lesions at electrode sites, uncontrolled epilepsy or history of seizure in the past 12 months
* Unstable medical or psychiatric conditions that preclude safe participation (e.g., uncontrolled hypertension, recent cardiovascular events, severe orthostatic hypotension with syncope)
* Severe freezing of gait or fall risk that prevents safe participation in supervised Nordic Walking, as judged by the clinical team
* Severe musculoskeletal or vestibular disorders that limit walking with poles; severe uncorrected visual impairment
* Cognitive impairment incompatible with consent or testing (e.g., MMSE <24)
* Current participation in other interventional trials targeting gait/balance or brain stimulation; recent initiation or dose change of antiparkinsonian medication within 4 weeks.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Gait speed (m/s) on the 10-Meter Walk Test (10MWT) | Baseline; Post-intervention (4 weeks); 1-month follow-up
  Preferred-pace 10MWT on a straight walkway with flying start; speed computed as distance/time (central 10 m if applicable), averaged across ≥2 trials. Higher values indicate better performance. The primary endpoint is the post-intervention assessment; maintenance is examined at 1 month. Minimally important change will be reported for clinical relevance.

SECONDARY OUTCOMES:
Timed Up and Go (seconds) | Baseline; Post-intervention; 1-month follow-up
  Time to stand up from a chair, walk 3 m, turn, return, and sit. Lower values indicate better performance.
Berg Balance Scale (0-56) | Baseline; Post-intervention; 1-month follow-up
  14-item balance assessment scored 0-4 each; total 0-56. Higher scores indicate better balance.
Freezing of Gait Questionnaire (FOG-Q; 0-24) | Baseline; Post-intervention; 1-month follow-up
  Patient-reported freezing severity/frequency. Higher scores indicate worse freezing.
MDS-UPDRS Part III - Motor Examination (0-132) | Baseline; Post-intervention; 1-month follow-up
  Clinician-rated motor signs of PD. Higher scores indicate greater impairment.
PDQ-39 Summary Index | Baseline; Post-intervention; 1-month follow-up
  Disease-specific quality of life; transformed 0-100%. Higher values indicate worse quality of life.
Adverse events related to tDCS and Nordic Walking (count and severity) | From first intervention session through 1-month follow-up
  Session-by-session standardized checklist for expected tDCS sensations (e.g., tingling, itching, erythema, headache, dizziness) and exercise-related symptoms; classification by severity and relatedness; serious adverse events recorded and reported per policy.
Step length during walking (meters) | Baseline; Post-intervention (4 weeks); 1-month follow-up
  Mean step length (m) at preferred walking speed on a straight walkway, averaged across ≥2 trials. Higher values indicate improvement.
Cadence during walking (steps/min) | Baseline; Post-intervention (4 weeks); 1-month follow-up
  Mean cadence (steps/min) at preferred walking speed on a straight walkway, averaged across ≥2 trials. Appropriate increases indicate improved gait rhythm.

CONTACTS AND LOCATIONS:
Locations (1):
- UEAFTO - Unidade de Fisioterapia e Terapia Ocupacional, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Undecided